CLINICAL TRIAL: NCT05920616
Title: Comprehensive Imaging Exam of Convalesced COVID-19 Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Canon Medical Systems, USA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00252436
Record Dates: First submitted 2023-06-23; First posted 2023-06-27 (Actual); Last update posted 2025-06-16 (Actual); Status verified 2025-06

CONDITIONS: COVID-19; COVID Long-Haul
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospitalized (Other): Participants who were hospitalized due to their COVID-19 illness.
  Interventions: Other: Magnetic Resonance Imaging; Other: Ultra-High Resolution Computed Tomography (CT) Scan
- Non-Hospitalized (Other): Participants who had COVID-19 but did not require hospitalization secondary to their illness.
  Interventions: Other: Magnetic Resonance Imaging; Other: Ultra-High Resolution Computed Tomography (CT) Scan

INTERVENTIONS:
Other: Magnetic Resonance Imaging — Completion of Magnetic Resonance Imaging of the brain, heart, lungs, and liver with and without contrast.
Other: Ultra-High Resolution Computed Tomography (CT) Scan — Completion of a high resolution CT scan of the lungs and high resolution CT of the coronary arteries.

SUMMARY:
COVID-19 is a systemic inflammatory disease involving many organs including the lungs, vascular system liver and myocardium that lead to severe pathologies. Patients with severe cardiopulmonary symptoms usually require weeks to months to fully recover. Studies of clinical and subclinical impairments of COVID-19 patients are important for medical practice and public health as well as providing pathogenic insight to the viral infection and secondary immune response. Chronic damage of vital organs and systems, and the potential long-term effects is of serious concern. In this study the investigators plan to quantify and characterize chronic consequences of COVID-19 in individuals who receive similar medical care related to disease severity and duration in a single health care system. Using state-of-the-art Computed Tomography (CT) and Magnetic Resonance Imaging (MRI) technology, we will study the pathology in major organ systems in comparison to matched controls. The results of this study may facilitate measures to prevent, detect, and manage complications from COVID-19 infections.

DETAILED DESCRIPTION:
As the number of recovered COVID-19 patients increase around the globe, it is important to understand the longterm impact of the disease so that healthcare systems and providers can optimize follow-up care of these patients. Identifying long term effects may also help identify patients with an increased risk of major adverse events following discharge from the hospital. Currently, the long term effects of COVID-19 in discharged hospitalized patients remain unknown. Infection with COVID-19 may result in involvement of many organ systems, including the lung, heart, brain, liver, and kidneys. Patients with a previous history of cardiovascular disease have been found to be at higher risk for incident cardiovascular complications. Direct or indirect effects of COVID-19 infection may predispose patients to thrombotic events including acute myocardial injury or pulmonary defects. Cardio-pulmonary features of COVID-19 include: bilateral multilobar ground-glass opacifications, septal thickening, bronchiectasis, pleural thickening, and subpleural involvement. Gradual resolution of consolidative opacities and other imaging patterns associated with clinical improvement usually occur after the second week of the disease. Characterization and quantification of organ injury as well associated organ dysfunction may help facilitating appropriate prevention and management.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18+
* Diagnosed with COVID-19 at any point starting March 2020.
* Subgroup A: hospitalized due to COVID-19 infection
* Subgroup B: non-hospitalized

Exclusion Criteria:

* Known allergy to either gadolinium or iodine based contrast agents
* Glomerular Filtration Rate (GFR) <45 mL/min (using the Cockcroft-Gault formula)
* Pregnancy
* Internal electrical devices, such as cochlear implant, spinal cord stimulator, pacemaker, or defibrillator
* Atrial fibrillation, uncontrolled tachyarrhythmia or advanced atrioventricular block (2nd or 3rd degree) at time of imaging
* Evidence of severe symptomatic heart failure (NYHA Class III or IV) at the time of imaging
* Other acute illness
* Ongoing mechanical ventilation related to hospitalization for COVID-19 related illness
* Presence of any other history or condition that the investigator feels would be problematic
* Weight exceeding 300 lbs (MRI table weight restrictions)
* Severe claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Degree and extent of fibrosis | Analyzed within 6 months of study completion
  - MRI to assess degree and extent of fibrosis in the liver, lungs, brain, myocardium, and vascular systems

SECONDARY OUTCOMES:
Assessment of Perfusion | Analyzed within 6 months of study completion
  Ultra-High Resolution CT to assess the amount of perfusion to the lungs and heart.

CONTACTS AND LOCATIONS:
Overall Officials: Joao Lima, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may provided to qualified researchers with academic interest in COVID-19. Data shared will not contain any personal health information (PHI). A statement of work and data use agreement are pre-requisites for data sharing.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 12 months after article publication. Data will be made accessible up to 24 months with extensions considered as needed.
Access Criteria: Access provided upon request.